CLINICAL TRIAL: NCT01292395
Title: The Musculoskeletal Response to Energy Deficit: Defining Optimal Protein Intake
Brief Title: Effects of Dietary Protein on Musculoskeletal Health During Calorie Deficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Army Research Institute of Environmental Medicine (U.S. Federal Agency)
Collaborators: USDA Grand Forks Human Nutrition Research Center (U.S. Federal Agency); Eastern Michigan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: H10-03; 503 (Other: USDA GFHNRC)
Record Dates: First submitted 2011-01-19; First posted 2011-02-09 (Estimated); Last update posted 2017-08-14 (Actual); Status verified 2017-08

CONDITIONS: Weight Loss; Muscle Loss; Bone Loss
Keywords: dietary supplement; protein metabolism; bone turnover
MeSH Terms: conditions — Weight Loss; Muscular Atrophy; Bone Diseases, Metabolic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Protein level 1 (Experimental)
  Interventions: Other: Dietary Protein Intake
- Protein level 2 (Experimental)
  Interventions: Other: Dietary Protein Intake
- Protein level 3 (Experimental)
  Interventions: Other: Dietary Protein Intake

INTERVENTIONS:
Other: Dietary Protein Intake — Protein intakes within the current recommendation

SUMMARY:
Military personnel face many physiological challenges, including sustained physical activity and prolonged periods of negative energy balance. Chronic energy deficiency often results in a loss of skeletal muscle mass and can reduce overall bone health. Recent evidence suggests that dietary interventions that provide protein in excess of the current national dietary recommendation may confer protection against the negative effects of energy deficiency on the musculoskeletal system. The primary objective of this randomized, controlled study is to assess the effects dietary protein intake spanning the current acceptable macronutrient distribution range on musculoskeletal health following prolonged energy deficiency. Findings from this investigation will improve current understanding of dietary conditions necessary to reduce the damaging effects of caloric deficiency on musculoskeletal health in warfighters. Furthermore, given the rise in obesity in military populations, findings may aid in the development of nutritional weight management strategies that promote healthy weight loss without compromising musculoskeletal health.

ELIGIBILITY:
Inclusion Criteria:

* Weight stable with body mass index 22-29 kg/m2
* Physically active
* Refrain from NSAIDS and other aspirin containing medications
* Refrain from alcohol and nicotine

Exclusion Criteria:

* Metabolic or cardiovascular abnormalities, gastrointestinal disorders
* Disease or medication that affects metabolism and/or exercise
* Allergies or intolerance to foods, vegetarian practices, or medications to be used in the study
* Anemia and Sickle Cell Anemia/Trait; abnormal PT/PTT test or problems with blood clotting
* Present condition of alcoholism, use of nutritional/sports supplements, anabolic steroids, or other substance abuse issues
* Musculoskeletal injuries that compromise the ability to exercise
* Blood donation within 8 weeks of beginning the study
* Pregnancy and women not on contraceptives

Ages: 18 Years to 42 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2010-09; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Change from weight maintenance in muscle metabolism after energy restriction | Measured after a 3 week energy deficit

SECONDARY OUTCOMES:
Change from weight maintenance in bone metabolism after energy restriction | Measured after a 3 week energy deficit

CONTACTS AND LOCATIONS:
Overall Officials: Stefan M Pasiakos, PhD, Principal Investigator — United States Army Research Institute of Environmental Medicine
Locations (1):
- USDA Grand Forks Human Nutrition Research Center, Grand Forks, North Dakota, United States

REFERENCES:
- [Background] Carbone JW, McClung JP, Pasiakos SM. Skeletal muscle responses to negative energy balance: effects of dietary protein. Adv Nutr. 2012 Mar 1;3(2):119-26. doi: 10.3945/an.111.001792. PMID 22516719
- [Result] Cao JJ, Pasiakos SM, Margolis LM, Sauter ER, Whigham LD, McClung JP, Young AJ, Combs GF Jr. Calcium homeostasis and bone metabolic responses to high-protein diets during energy deficit in healthy young adults: a randomized controlled trial. Am J Clin Nutr. 2014 Feb;99(2):400-7. doi: 10.3945/ajcn.113.073809. Epub 2013 Nov 27. PMID 24284444
- [Result] Pasiakos SM, Margolis LM, McClung JP, Cao JJ, Whigham LD, Combs GF, Young AJ. Whole-body protein turnover response to short-term high-protein diets during weight loss: a randomized controlled trial. Int J Obes (Lond). 2014 Jul;38(7):1015-8. doi: 10.1038/ijo.2013.197. Epub 2013 Oct 29. PMID 24166063
- [Result] Carbone JW, Margolis LM, McClung JP, Cao JJ, Murphy NE, Sauter ER, Combs GF Jr, Young AJ, Pasiakos SM. Effects of energy deficit, dietary protein, and feeding on intracellular regulators of skeletal muscle proteolysis. FASEB J. 2013 Dec;27(12):5104-11. doi: 10.1096/fj.13-239228. Epub 2013 Aug 21. PMID 23965841
- [Result] Pasiakos SM, Cao JJ, Margolis LM, Sauter ER, Whigham LD, McClung JP, Rood JC, Carbone JW, Combs GF Jr, Young AJ. Effects of high-protein diets on fat-free mass and muscle protein synthesis following weight loss: a randomized controlled trial. FASEB J. 2013 Sep;27(9):3837-47. doi: 10.1096/fj.13-230227. Epub 2013 Jun 5. PMID 23739654
- [Derived] Karl JP, Thompson LA, Niro PJ, Margolis LM, McClung JP, Cao JJ, Whigham LD, Combs GF Jr, Young AJ, Lieberman HR, Pasiakos SM. Transient decrements in mood during energy deficit are independent of dietary protein-to-carbohydrate ratio. Physiol Behav. 2015 Feb;139:524-31. doi: 10.1016/j.physbeh.2014.11.068. Epub 2014 Dec 3. PMID 25479571
- [Derived] Henning PC, Margolis LM, McClung JP, Young AJ, Pasiakos SM. High protein diets do not attenuate decrements in testosterone and IGF-I during energy deficit. Metabolism. 2014 May;63(5):628-32. doi: 10.1016/j.metabol.2014.02.007. Epub 2014 Feb 17. PMID 24641883